CLINICAL TRIAL: NCT05939687
Title: Prophylactic Mesh Placement During Temporary Stoma Closure: a Prospective Randomized Phase III Clinical Trial
Brief Title: Prophylactic Mesh Placement During Stoma Closure After Low Anterior Resection
Acronym: ProMeLAR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Principal Investigator, Sergey Gordeyev, Principal investigator, Department of Colorectal surgery, Blokhin's Russian Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ProMeLAR-01
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Neoplasms Malignant; Rectal Cancer; Hernia Incisional; Surgery
Keywords: Rectal cancer; mesh; stoma-site hernia; prevention; surgery
MeSH Terms: conditions — Neoplasms; Rectal Neoplasms; Incisional Hernia | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Intervention Model Description: 1:1 electronic randomisation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mesh (Experimental): In these patients we will do sublay/interoblique repair for prevention of stoma-site hernias using a polypropylene mesh.
  Interventions: Procedure: mesh
- non-mesh (Active Comparator): In these patients we will close the stoma with standard layered ligature suturing of the abdominal wall without mesh implantation.
  Interventions: Procedure: non-mesh

INTERVENTIONS:
Procedure: mesh — We'll use mesh repair for prevention of stoma-site hernias in the study group.
  Other Names: polypropylene mesh
  Arms: mesh
Procedure: non-mesh — We'll use the layered ligature suturing of the abdominal wall without mesh implantation in the control group.
  Arms: non-mesh

SUMMARY:
The goal of this clinical trial is to compare the efficacy of using polypropylene mesh for hernia prevention after stoma closure in patients with colorectal cancer and non-mesh repair. The main question it aims to answer is: can mesh help prevent hernia? Participants will be divided into 2 groups: with and without mesh using. They must be followed up for 2 years after enrollment in the study.

Researchers will compare mesh and non-mesh groups to evaluate the benefits and harms of mesh using in hernia prevention.

DETAILED DESCRIPTION:
This clinical trial is prospective randomized phase III study of the efficacy of polypropylene mesh for hernia prevention after stoma closure in patients with colorectal cancer. We will include in the study group 71 patients with colorectal cancer with ileo- and colostomy. In these patients we will do sublay/interoblique repair in prevention incisional hernias using polypropylene mesh. Our hypothesis is to reduce parastomal hernias rate from 30% to 10% over 2 years. Stratification will be used for patients with >5 cm vs <5 cm stoma-site hernia.

The control group will include 71 patients with similar parameters who will undergo stoma closure with layered ligature suturing of the abdominal wall without mesh implantation.

Additional endpoints are the wound infection rate, the complication rate (Clavien-Dindo), the rate of the repeated surgery for hernia at the site of stoma closure. We'll assess the quality of life by HerQLes (Hernia-Related Quality of Life Survey) scale.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Absence of distant metastases (M0)
* ECOG (Eastern Cooperative Oncology Group) status 0-2
* completed course of adjuvant treatment
* Absence of acute inflammatory parastomal complications
* Integrity of colorectal anastomosis

Exclusion Criteria:

* Inability to obtain consent to participate
* Synchronous and metachronous malignant neoplasms
* Clinically significant diseases of the cardiovascular system, liver, kidney, central nervous system
* Parastomal inflammation and other conditions that increase the risk of postoperative complications
* Pregnancy
* HIV infection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
hernia rate | 2 years
  The rate of parastomal hernias after stoma closure for 2 years.

SECONDARY OUTCOMES:
90 day surgical morbidity | 90 days
  Complications after stoma closure including hernias
Quality of life indicators by HerQLes scale | 2 years
  Quality of life as assessed by Hernia-Related Quality of Life Survey scale (HerQLes) at 30 days, 1 year and 2 years after stoma closure (higher scores are worse)

CONTACTS AND LOCATIONS:
Overall Officials: Zaman Z Mamedli, PhD, Study Director — N.N.Blokhin Russian Cancer Research Center; Nikolay L Matveev, PhD, Study Chair — Pirogov Russian National Research Medical University
Locations (1):
- N.N.Blokhin Russian Cancer Research Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No